CLINICAL TRIAL: NCT00699855
Title: Observational Long-term Follow-up of the Phase IV Open-label Trial of Predictive Markers in GHD and TS Pre-pubertal Children Treated With Saizen
Brief Title: Long Term Follow up Study of Predictive Markers in GHD and TS Children
Acronym: PREDICT LT FUP
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Other Study IDs: 28614
Record Dates: First submitted 2008-06-13; First posted 2008-06-18 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Growth Hormon Deficiency; Turner Syndrome in Pre-pubertal Children
Keywords: Growth Hormon Deficiency and; Turner Syndrome in pre-pubertal children; Long term follow-up of predictive markers

SUMMARY:
Primary objective is to assess the relationship between changes from serum biomarkers observed after 1 month of Saizen® therapy and change in height, weight after up to 5 years of treatment with Growth Hormone in children with Growth Hormone Deficiency (GHD) and Turner Syndrome (TS).

DETAILED DESCRIPTION:
This study is an observational study that will collect data from patients enrolled in a previous study (PREDICT, NCT 00256126). Data such as auxological parameters (height, weight, Tanner stage, bone age will be collected as well as GH treatment use (including dose and adherence to the treatment).

Because for some countries the start of this long term follow up study will take place more than one year after subjects have completed the initial study (PREDICT) retrospective data may be collected (if subjects agree) as well as prospective data.

When available laboratory parameters such as IGF-1, IGFPB-3, fasting glucose, fasting insulin, TSH and T4 will also be collected.

This data will be collected yearly during the normal follow up visits during 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Have completed the PREDICT study (NCT 00256126)
* Followed up at least 1 year when still under treatment after completion of PREDICT Trial
* Parent's or guardian's written consent given before any data collection

Exclusion Criteria:

* Use of an investigational drug or participation in another interventional clinical trial since discontinuation of PREDICT trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects initially enrolled in PREDICT (NCT 00256126) clinical study and continuing a growth hormone treatment.
Sampling Method: Non-Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2008-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Data such as auxological parameters (height, weight, Tanner stage, bone age) will be collected as well as GH treatment use (including dose and adherence to the treatment). | Yearly

SECONDARY OUTCOMES:
When available laboratory parameters such as IGF-1, IGFPB-3, fasting glucose, fasting insulin, TSH and T4 will also be collected. | Yearly

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Della Corte, Study Director — Merck Serono S.A., Geneva

REFERENCES:
- [Result] Clayton P, Chatelain P, Tato L, Yoo HW, Ambler GR, Belgorosky A, Quinteiro S, Deal C, Stevens A, Raelson J, Croteau P, Destenaves B, Olivier C. A pharmacogenomic approach to the treatment of children with GH deficiency or Turner syndrome. Eur J Endocrinol. 2013 Jul 29;169(3):277-89. doi: 10.1530/EJE-13-0069. Print 2013 Sep. PMID 23761422
- [Derived] Stevens A, Murray P, De Leonibus C, Garner T, Koledova E, Ambler G, Kapelari K, Binder G, Maghnie M, Zucchini S, Bashnina E, Skorodok J, Yeste D, Belgorosky A, Siguero JL, Coutant R, Vangsoy-Hansen E, Hagenas L, Dahlgren J, Deal C, Chatelain P, Clayton P. Gene expression signatures predict response to therapy with growth hormone. Pharmacogenomics J. 2021 Oct;21(5):594-607. doi: 10.1038/s41397-021-00237-5. Epub 2021 May 27. PMID 34045667
- [Derived] Murray PG, Stevens A, De Leonibus C, Koledova E, Chatelain P, Clayton PE. Transcriptomics and machine learning predict diagnosis and severity of growth hormone deficiency. JCI Insight. 2018 Apr 5;3(7):e93247. doi: 10.1172/jci.insight.93247. eCollection 2018 Apr 5. PMID 29618660
- [Derived] De Leonibus C, Chatelain P, Knight C, Clayton P, Stevens A. Effect of summer daylight exposure and genetic background on growth in growth hormone-deficient children. Pharmacogenomics J. 2016 Nov;16(6):540-550. doi: 10.1038/tpj.2015.67. Epub 2015 Oct 27. PMID 26503811
- [Derived] Valsesia A, Chatelain P, Stevens A, Peterkova VA, Belgorosky A, Maghnie M, Antoniazzi F, Koledova E, Wojcik J, Farmer P, Destenaves B, Clayton P; PREDICT Investigator group. GH deficiency status combined with GH receptor polymorphism affects response to GH in children. Eur J Endocrinol. 2015 Dec;173(6):777-89. doi: 10.1530/EJE-15-0474. Epub 2015 Sep 4. PMID 26340968